CLINICAL TRIAL: NCT07285343
Title: Controlled Randomized Clinical Trial of Containment of the Elevator Muscle of Upper Lip and Wing of Nose Technique Versus Conventional Lip Repositioning for Treatment of Gummy Smile
Brief Title: Comparison Between Lip Repositioning and Muscle Traction Technique in Treatment of Gummy Smile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 240/2019 suez canal university
Record Dates: First submitted 2025-09-22; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-09

CONDITIONS: Gummy Smile Due to Hypermobile Upper Lip; Excessive Gingival Display
Keywords: Gummy Smile; Patient Discomfort; Patient Satisfaction; Gingival Display; Smile Line; Smile index; lip repositioning; muscle traction
MeSH Terms: conditions — Patient Satisfaction | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single-blinded technique
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lip repositioning (Active Comparator): lip repositioning to treat excessive gingival display
  Interventions: Procedure: lip repositioning
- Containment of the elevator muscle of the upper lip and wing of nose (EMULWN) (Active Comparator): Containment of the elevator muscle of the upper lip and wing of nose (EMULWN) technique in treatment of excessive gingival display
  Interventions: Procedure: Containment of the elevator muscle of the upper lip and wing of nose (EMULWN) technique

INTERVENTIONS:
Procedure: lip repositioning — Local anesthesia was administered in the vestibular mucosa. A partial-thickness incision was made at the mucogingival junction from the mesial line angle of the right first molar to the mesial line angle of the left first molar. A second partial- thickness incision, parallel to the first, was made in the labial mucosa, 10 to 12 mm apical to the mucogingival junction. The incisions were connected at each first molar, creating an elliptical outline. The epithelium was removed within the outline of the incisions, leaving the underlying connective tissue exposed. Care was taken to avoid damage to any minor salivary glands in the submucosa. The parallel incision lines were approximated with interrupted stabilization sutures at the midline and other locations along the borders of the incision to ensure proper alignment of the lip midline with the midline of the teeth. Then, a continuous interlocking suture was used to approximate both flap ends.
  Arms: lip repositioning
Procedure: Containment of the elevator muscle of the upper lip and wing of nose (EMULWN) technique — Local anesthesia was administered in the vestibular mucosa and lip then a vertical incision was made on the labial frenum, and two more horizontal incisions were made on the mucogingival line, starting from the frenum incision up to the height of the canines. The flap was carefully divulsed with Goldman Fox scissors and also a curved hemostat, separating the external epithelium from the muscle bundle mucosa on both sides at the height of the lateral incisors and canines. With an absorbable suture thread, the elevator muscle of the upper lip and wing of the nose was pulled downwards, repositioning its bundle nearer the highest portion of the keratinized gingiva. Simple sutures were made, as many as necessary, in order to contain the pulled muscle in this position. The procedure ended up with a continuous suture in the labial frenum and in the horizontal incisions with the use of a 4-0 silk suture thread. The external stitches should be removed in 10-15 days" time.
  Arms: Containment of the elevator muscle of the upper lip and wing of nose (EMULWN)

SUMMARY:
The goal of this clinical trial is to compare and evaluate the effectiveness of conventional and modified lip repositioning for the treatment of gummy smile.

The main question it aims to answer:

Which of these treatment modalities (conventional lip repositioning and containment of the elevator muscle of the upper lip and wing of nose (EMULWN)) has the most durable and least relapse in the treatment of gummy smile?"

Researchers will compare:

1. The primary outcome was the decrease in excessive gingival display by measuring smile line (gingival display) and smile index before and after treatment modalities.
2. The The secondary outcome was to measure the durability and possibility of relapse over 6 months after treatment with high patient satisfaction.

DETAILED DESCRIPTION:
For patients seeking long-term correction of excessive gingival displays, there are different treatment modalities. Both lip repositioning and muscle traction techniques showed improvement in the decrease in the amount of gingival display, while the containment surgery of the muscle of the upper lip and wing of the nose showed durable and satisfactory esthetics with less patient discomfort and less pain immediately after the procedure and needs more time to study or may need some modification. Also, lip repositioning showed satisfactory results to the patients but with more pain immediately after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged between 18 and 38 years.
2. Gummy smile ranging between 4 and 6 mm, due to short upper lip and hyperactive lip elevator muscles (lip mobility >8 mm).
3. Good periodontal health based on the examination of the gingival inflammation index, bleeding index, and probing the depth of gingival pockets.
4. Healthy patients or people with well-controlled systemic disease.

Exclusion Criteria:

1. Smokers.
2. Pregnant or lactating women.
3. Less than 3 mm of attached gingiva that might create difficulties in flap design, stabilization, and suturing.
4. Vertical maxillary excess of more than 6 mm.
5. Poorly controlled systemic diseases that preclude local anesthesia.
6. Altered passive eruption, which needs gingivectomy or an apically positioned flap.
7. Skeletal causes of gummy smile as protruded maxilla.

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Measuring smile line (the amount of gingival display in millimeters) | at baseline, after one month, after 3 months and after 6 months
  The first primary outcome of the study was to measure the change in excessive gingival display by measuring smile line (the amount of gingival display in millimeters) before and after treatment.
  1/Smile line (gingival display) Type 1: Very high smile line: 2 mm or more of marginal and attached gingiva visible or more than 2 mm of root or gingiva apical to the cemento-enamel junction visible for the healthy but reduced periodontium. This smile is classified as a "gummy smile." Type 2: High smile line: Between 0 and 2 mm of marginal and attached gingiva visible or between 0 and 2 mm visibility of root and gingiva apical to the cemento-enamel junction visible for the reduced and healthy periodontium.
  Type 3: Average smile line: Gingival embrasures only visible. Type 4: Low smile line: Gingival embrasure and cemento-enamel junction not visible.
Measuring smile index ratio before and after treatment. | at baseline, after one month, after 3 months and after 6 months
  The second primary outcome of the study was to measure the change in excessive gingival display by measuring smile index ratio which is (intercommissural width/interlabial gap) to visualize and quantify the frontal smile. The ratio is used for comparing smiles among patients. The lower the smile index, the less youthful the smile appears.

SECONDARY OUTCOMES:
Patient Satisfaction with Their Smile | at baseline, one month, 3 months and 6 months
  Patient satisfaction with their smile was recorded on the following scale: 0 (very satisfied); 1 (satisfied); 2 (moderately satisfied); 3 (unsatisfied).
Patient discomfort | immediately after treatment
  Patient discomfort was recorded on a visual analog scale, with scores from 0 to 10, where 0 corresponds to no discomfort and 10 corresponds to maximum discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Hany Kamel Shalaby, professor, Principal Investigator — Suez Canal University
Locations (2):
- Egypt (2):
  - Periodontology Clinic in Suez Canal University, Cairo, Egypt
  - Periodontology Clinic in Suez Canal University, Ismailia, Ismailia Governorate

IPD SHARING:
Plan to Share IPD: No